CLINICAL TRIAL: NCT02985125
Title: A Phase I/II Study of LEE011 Plus Everolimus in Patients With Metastatic Pancreatic Adenocarcinoma Refractory to Chemotherapy
Brief Title: LEE011 Plus Everolimus in Patients With Metastatic Pancreatic Adenocarcinoma Refractory to Chemotherapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Georgetown University (Other)
Collaborators: Novartis (Industry); University of Texas Southwestern Medical Center (Other); Cedars-Sinai Medical Center (Other); Virginia Mason Hospital/Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0232
Record Dates: First submitted 2016-11-29; First posted 2016-12-07 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: Pancreas; 5-FU; Gemcitabine; LEE011; Everolimus; Refractory; Chemotherapy
MeSH Terms: interventions — ribociclib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase I - Dose Level 1 (Experimental): Treatment cycles are 28 days long.
  LEE011 (taken orally) - 250mg Once daily on days 1-21
  Everolimus (taken orally) - 2.5mg Once daily on days 1-28
  Interventions: Drug: LEE011; Drug: Everolimus
- Phase I - Dose Level 2 (Experimental): Treatment cycles are 28 days long.
  LEE011 (taken orally) - 300mg Once daily on days 1-21
  Everolimus (taken orally) - 2.5mg Once daily on days 1-28
  Interventions: Drug: LEE011; Drug: Everolimus
- Phase I - Dose Level -1 (Experimental): Treatment cycles are 28 days long.
  LEE011 (taken orally) - 200mg Once daily on days 1-21
  Everolimus (taken orally) - 2.5mg Once daily on days 1-28
  Interventions: Drug: LEE011; Drug: Everolimus
- Phase I - Dose Level -2 (Experimental): Treatment cycles are 28 days long.
  LEE011 (taken orally) - 150mg Once daily on days 1-21
  Everolimus (taken orally) - 2.5mg Once daily on days 1-28
  Interventions: Drug: LEE011; Drug: Everolimus
- Phase II - Dose (Experimental): Treatment cycles are 28 days long.
  LEE011 (taken orally) - the recommended phase II dose Once daily on days 1-21
  Everolimus (taken orally) - 2.5mg Once daily on days 1-28
  Interventions: Drug: LEE011; Drug: Everolimus

INTERVENTIONS:
Drug: LEE011 — Treatment cycles are 28 days long. It is taken orally. The dosage varies depending on the study arm.
  Other Names: ribociclib
Drug: Everolimus — Treatment cycles are 28 days long. It is taken orally. On all arms, the dosage will be 2.5mg.
  Other Names: Afinitor®

SUMMARY:
This study is a single-arm, open-label, multi-institutional Phase I/II trial of the combination of LEE011 and everolimus in refractory mPAC.

DETAILED DESCRIPTION:
This is a single arm, open label Phase I/II study to evaluate the progression free survival at 8 weeks (PFS8week) of the combination of LEE-011 plus everolimus, in patients with metastatic pancreatic cancer refractory to 5-fluorouracil (5-FU) and gemcitabine-based chemotherapy. Previous studies of third-line therapy in mPAC are limited but reveal stable disease in 25-31% of patients with no partial or complete responses (31% of patients in the GVAX/CRS-207 combination vaccine study had stable disease but only 52% of these patients were treated in the third-line setting). It is hoped that the combination of LEE-011 plus everolimus can increase the PFS8weeks to at least 50%, though early stopping rules are in place for lack of efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed mPAC (mixed histology is acceptable as long as the predominant histology is pancreatic adenocarcinoma)
2. Patient must consent to two mandatory biopsies and have tumor amenable to biopsy
3. Measurable disease by RECIST v1.1 criteria (tumor ≥ 1 cm in longest diameter on axial image on CT or MRI and/or lymph node(s) ≥ 1.5 cm in short axis on CT or MRI) on baseline imaging
4. Documented progression of disease on at least one 5-FU-based regimen and at least one GEM-based regimen for metastatic disease (progression during or within 3 months of the completion of adjuvant therapy is acceptable)
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2 (see Table 2)
6. Age ≥ 18 years
7. Subjects with no brain metastases or a history of previously treated brain metastases who have been treated by surgery or stereotactic radiosurgery (SRS) at least 4 weeks prior to enrollment and have a baseline MRI that shows no evidence of active intracranial disease
8. Patients with available standard 12-lead ECG with the following parameters at screening (defined as the mean of the triplicate ECGs):

   * QTcF interval at screening <450msec
   * Resting heart rate 50-90bpm
9. Bone marrow function: absolute neutrophil count (ANC) ≥ 1,500/mm3; Platelets ≥100 × 109/L; hemoglobin ≥ 9.0 g/dL

   • Patients may have a transfusion of red blood cells to meet the hemoglobin requirement
10. Renal function: serum creatinine ≤ 1.5 × upper normal limit of institution's normal range or creatinine clearance ≥ 50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal
11. Hepatic function: Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3.0 × the upper normal limit of institution's normal range. Total bilirubin ≤ 1.5 × the upper normal limit of institution's normal range. For subjects with liver metastases, AST and ALT < 5 × the upper normal limit of institution's normal range, and total bilirubin >1.5 - 3.0 x the upper normal limit of institution's normal range are acceptable as long as there is no persistent nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia.
12. Partial Thromboplastin Time (PTT) must be ≤ 1.5 × upper normal limit of institution's normal range and International Normalized Ratio (INR) < 1.5. Subjects on anticoagulant (such as warfarin) will be permitted to enroll as long s the INR is in the acceptable therapeutic range as determined by the investigator.
13. Potassium, total calcium (corrected for serum albumin), magnesium, sodium and phosphorus within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication
14. Patients must have fully recovered from all effects of surgery. Patients must have had at least two weeks after minor surgery and four weeks after major surgery before starting therapy. Minor procedures requiring "Twilight" sedation such as endoscopies or mediport placement may only require a 24-hour waiting period, but this must be discussed with an investigator.
15. Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to initiation of treatment and/or postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential
16. Patient is capable of swallowing pills whole
17. Patient is capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consent, approved by the Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures

Exclusion Criteria:

1. Patients previously exposed to, intolerant of, or ineligible for Cyclin-dependent kinase (CDK) inhibitors, Mammalian target of rapamycin (mTOR) inhibitors, and/or their combination
2. Prior anti-tumor therapy within 3 weeks of Cycle 1 Day 1 (anti-tumor therapy defined as, but is not limited to, anti-cancer agents (cytotoxic chemotherapy, immunotherapy, and biologic therapy), radiotherapy, and investigational agents), the "wash-out period"
3. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.).
4. Women who are pregnant or breastfeeding
5. Concurrent use of CYP3A4 inhibiting or activating medications
6. Concurrent use of an Angiotensin-converting enzyme (ACE) inhibitor (increased risk of angioedema with ACE inhibitors administered in combination with everolimus, seen in approximately 6.8% of patients)
7. Psychiatric illness or social situation that would limit compliance with study requirements
8. Patient has a concurrent malignancy or malignancy within 3 years prior to starting study drug, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer.
9. Patients with central nervous system (CNS) involvement unless they meet ALL of the following criteria:

   * At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment
   * Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases.
10. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
11. Patient has a known history of HIV infection or chronic, active Hepatitis B (testing not mandatory).
12. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.).
13. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormalities, including any of the following:

    * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to screening
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
    * Documented cardiomyopathy
    * Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening
    * Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade Atrioventricular block (AV) block (e.g. bifascicular block, Mobitz type II and third-degree AV block)
    * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:
    * Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
    * Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued (within 5 half-lives or 7 days prior to starting study drug) or replaced by safe alternative medication
    * Inability to determine the QT interval on screening (QTcF, using Fridericia's correction)
    * Systolic blood pressure (SBP) >160 mmHg or <90 mmHg at screening
14. Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to starting study drug (see Table 4 for details):

    * Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges
    * That have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
    * Herbal preparations/medications, dietary supplements.
15. Patient is currently receiving or has received systemic corticosteroids ≤2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-05-04 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate at 8 weeks | 8 weeks
  PFS at 8 weeks in a patient with refractory mPAC treated with LEE011 and everolimus, defined as positive if a patient does not have evidence of progressive disease at 8 weeks as measured by expert radiologists using RECIST v1.1 criteria

SECONDARY OUTCOMES:
Progression-free survival | 2 years
  PFS in a patient with refractory mPAC treated with LEE011 and everolimus, defined as the time from Cycle 1, Day 1 to progressive disease (as measured by expert radiologists using RECIST v1.1 criteria), death from any cause, or last follow-up, as determined by the investigator of LEE011 and everolimus in patients with mPAC refractory to chemotherapy
Overall survival (OS) | 2 years
  Overall survival (OS) in a patient with refractory mPAC treated with LEE011 and everolimus, defined as the time from Cycle 1, Day 1 to death from any cause or last follow-up
Best response in a patient using RECIST v1.1 criteria | 2 years
  Best response in a patient, defined as the largest percent decrease in tumor size from baseline and categorized as a complete response, partial response, or stable disease by imaging studies, measured by expert radiologists using RECIST v1.1 criteria
Number of adverse events as accessed by NCI CTCAE v4.03 | 2 years
  Adverse events in a patient with refractory mPAC treated with LEE011 and everolimus, defined as the number of grade 3 and 4 toxicities according to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE v4.03) that occur after Cycle 1, Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Weinberg, MD, Study Chair — Lombardi Comprehensive Cancer Center
Locations (1):
- Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No